CLINICAL TRIAL: NCT04180228
Title: Human Papilloma Virus Vaccination and Chronic Inflammatory Rheumatic Disease. A Cross-sectional Study of Vaccinal Coverage, Barriers and Motivations.
Brief Title: Human Papilloma Virus Vaccination and Chronic Inflammatory Rheumatic Diseases.
Acronym: HPV-CIR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0456
Record Dates: First submitted 2019-10-31; First posted 2019-11-27 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Systemic Lupus Erythematosus; Idiopathic Juvenile Arthritis; Human Papilloma Virus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic lupus erythematosus: Investigators include in this group all young girls between 11 to 19 years old who accepted to respond to the questionnaire with systemic lupus erythematosus.
  Interventions: Other: self-administred questionnaire
- Idiopathic juvenile arthritis: Investigators include in this group all young girls between 11 to 19 years old who accepted to respond to the questionnaire, with idiopathic juvenile arthritis.
  Interventions: Other: self-administred questionnaire

INTERVENTIONS:
Other: self-administred questionnaire — On the occasion of a follow-up consultation with referent pediatrician, a self-administred questionnaire is distributed. It will take around ten minutes to the patient and her parents for completing the questionnaire. Questionnaire is anonymous. Participation is free and informed by an information notice. There is a list of items to complete by the patient and her parents. Most of questions are closed-ended. Clinical data are reported : age, level of education, principal disease (SLE or Juvenile arthritis), received treatments. In the questionnaire, it is asked if the patient is vaccinated or not for HPV, and reasons for it.

SUMMARY:
Patients with chronic inflammatory rheumatic disease (CIR) are at increased risk for infections. Vaccination is a powerful tool to prevent infections, even in immunocompromised patients. Low-risk types of Human papilloma virus (HPV) cause anogenital warts, while high risk types are strongly related to pre-malignant cervical abnormalities and cervical cancer. HPV vaccines have been developed to prevent these conditions. Human papillomavirus (HPV) infections are more prevalent in systemic lupus erythematosus (SLE) patients or other auto-immune diseases when compared to the healthy population. In France, despite a vaccination available since 2007, rate of vaccination remain low. Although little is known about HPV vaccination in SLE, few studies in patients with autoimmune rheumatic diseases (AIRDs) have shown that HPV vaccines are safe, and capable to induce an immunogenic response in this group of patients. To date, available data suggest that HPV vaccines can be given safely to SLE patients. Given the increased incidence of cervical abnormalities due to HPV in SLE patients, this vaccination should be encouraged.

The aim of this study was to assess the vaccination coverage rate in chronically ill girls with SLE or idiopathic juvenile arthritis who require a close pediatric specialized follow-up vaccination and to understand barriers or motivations for it.

ELIGIBILITY:
Inclusion Criteria:

* Young girls older than 11 years old until adult transition
* Follow-up for systemic lupus erythematosus (American college of rheumatology classification) or idiopathic juvenile arthritis (International League of Associations for Rheumatology classification)
* Follow-up in a Childen's hospital of Lyon (Hopital Femme Mère Enfant) and Paris (Hospital Necker-Enfants Malades, Hôpital Robert Debré)
* With no parental opposition to participate

Exclusion Criteria:

* Refusing to participate
* Age < 11 years old

Ages: 11 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Investigators study a French sample of young girls follow-up for systemic lupus erythematosus or idiopathic juvenile arthritis. It's a multicenter design.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Frequency of HPV vaccination (percentage of patients vaccinated). | Day 0, Time of intervention (questionnaire)
  We report this information with an item "vaccination for Human papilloma virus". The proposition of response is "Yes" or "No". We'll calculate the number of vaccination among the population including in the study.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Necke -, Enfants Malades, Paris
  - Service de médecine interne, Centre hospitalier Lyon Sud, Pierre-Bénite